CLINICAL TRIAL: NCT03190915
Title: A Phase 2 Study of the MEK Inhibitor Trametinib (NSC# 763093) in Children With Relapsed or Refractory Juvenile Myelomonocytic Leukemia
Brief Title: Trametinib in Treating Patients With Relapsed or Refractory Juvenile Myelomonocytic Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-00921; NCI-2017-00921 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ADVL1521 (Other: Children's Oncology Group); ADVL1521 (Other: CTEP); U10CA180886 (NIH); U54CA196519 (NIH)
Record Dates: First submitted 2017-06-16; First posted 2017-06-19 (Actual); Results first posted 2024-07-16 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-07

CONDITIONS: Juvenile Myelomonocytic Leukemia; Neurofibromatosis Type 1
MeSH Terms: conditions — Leukemia, Myelomonocytic, Juvenile; Neurofibromatosis 1 | interventions — Biopsy; trametinib; omipalisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (trametinib) (Experimental): Patients receive trametinib PO QD on days 1-28 of each cycle. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo a bone marrow aspiration or biopsy at baseline, on day 28 of cycles 1 and 2, at all subsequent odd numbered cycles, and at end of treatment.
  Interventions: Procedure: Bone Marrow Aspiration and Biopsy; Drug: Trametinib

INTERVENTIONS:
Procedure: Bone Marrow Aspiration and Biopsy — Undergo bone marrow aspiration or biopsy
Drug: Trametinib — Given PO
  Other Names: GSK 1120212; GSK 212; GSK-1120212; GSK-212; GSK1120212; GSK212; JTP 74057; JTP-74057; JTP74057; MEK Inhibitor GSK1120212

SUMMARY:
This phase II trial studies how well trametinib works in treating patients with juvenile myelomonocytic leukemia that has come back (relapsed) or does not respond to treatment (refractory). Trametinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the objective response rate to trametinib in children with recurrent or refractory juvenile myelomonocytic leukemia (JMML).

SECONDARY OBJECTIVES:

I. To further define and describe the toxicities of single agent trametinib in children with recurrent or refractory JMML.

II. To further characterize the pharmacokinetics of trametinib in children with recurrent or refractory JMML.

III. To prospectively evaluate mutant allele burden as a marker of disease activity in JMML.

IV. To measure the rate of complete responses in children with recurrent or refractory JMML.

V. To measure the duration of response among responders.

EXPLORATORY OBJECTIVE:

I. To describe the distribution of JMML diagnostic criteria in children with recurrent or refractory JMML.

OUTLINE:

Patients receive trametinib orally (PO) once daily (QD) on days 1-28 of each cycle. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo a bone marrow aspiration or biopsy at baseline, on day 28 of cycles 1 and 2, at all subsequent odd numbered cycles, and at end of treatment.

After completion of study treatment, patients are followed up annually for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be >= 1 month and < 22 years of age at the time of study entry
* Patients must have had histologic verification of juvenile myelomonocytic leukemia (JMML) at original diagnosis and currently have relapsed or refractory disease; the diagnosis is made based on the following criteria

  * JMML category 1 (all of the following): the diagnostic criteria must include all features in category 1 and EITHER (i) one of the features in category 2 OR (ii) two features from category 3 to make the diagnosis

    * Splenomegaly
    * > 1000 (1 x 10^9/uL) circulating monocytes
    * < 20% blasts in the bone marrow or peripheral blood
    * Absence of the t(9;22) or BCR/ABL fusion gene
  * JMML category 2 (at least one of the following if at least two category 3 criteria are not present):

    * Somatic mutation in RAS or PTPN11
    * Clinical diagnosis of NF1 or NF1 gene mutation
    * Homozygous mutation in CBL
    * Monosomy 7
  * JMML category 3 (at least two of the following if no category 2 criteria are met):

    * Circulating myeloid precursors
    * White blood cell count, > 10 000 (10 x 10^9/ uL)
    * Increased hemoglobin F for age
    * Clonal cytogenetic abnormality
    * GM-CSF hypersensitivity
* Patients with refractory or relapsed JMML must have had at least one cycle of intensive frontline therapy or at least 2 cycles of a deoxyribonucleic acid (DNA) demethylating agent with persistence of disease, defined by clinical symptoms or the presence of a clonal abnormality; frontline therapy is defined as one cycle of intravenous chemotherapy that includes any of the following agents: fludarabine, cytarabine, or any anthracycline but specifically excludes oral 6-mercaptopurine; frontline therapy will also include any conditioning regimen as part of a stem cell transplant; patients who transform to AML at any point with more than 20% blasts are not eligible for this trial
* Patients must have a Lansky or Karnofsky performance status score of >= 50, corresponding to Eastern Cooperative Oncology Group (ECOG) categories 0, 1 or 2; use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to study enrollment

  * Myelosuppressive chemotherapy: patients must have completely recovered from all acute toxic effects of chemotherapy, immunotherapy or radiotherapy prior to study enrollment; at least 14 days must have elapsed since the completion of cytotoxic therapy, with the exception of hydroxyurea

    * Note: cytoreduction with hydroxyurea can be initiated and continued for up to 24 hours prior to the start of protocol therapy
  * Hematopoietic growth factors: at least 14 days after the last dose of a long-acting growth factor (e.g., pegfilgrastim) or 7 days for short-acting growth factor; for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur
  * Biologic (anti-neoplastic agent): at least 7 days must have elapsed since completion of therapy with a biologic agent; for agents that have known adverse events occurring beyond 7 days after administration, this period prior to enrollment must be extended beyond the time during which adverse events are known to occur
  * Monoclonal antibodies:

    * At least 30 days after the completion of any type of immunotherapy, e.g. tumor vaccines
    * At least 3 half-lives must have elapsed since prior therapy that included a monoclonal antibody
  * Radiotherapy:

    * >= 2 weeks must have elapsed since local palliative external radiation therapy (XRT) (small port)
    * >= 6 months must have elapsed if prior craniospinal XRT was received, if >= 50% of the pelvis was irradiated, or if traumatic brain injury (TBI) was received
    * >= 4 weeks must have elapsed if other substantial bone marrow irradiation was given
  * Stem cell transplant or rescue without TBI: no evidence of active graft versus (vs.) host disease and >= 3 months must have elapsed since transplant; >= 4 weeks must have elapsed since any donor lymphocyte infusion
* Patients must not be known to be refractory to red blood cell or platelet transfusions
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 (within 7 days prior to enrollment) or a serum creatinine based on age/gender as follows (within 7 days prior to enrollment):

  * Age: Maximum serum creatinine (mg/dL)

    * 1 month to < 6 months: 0.4 (male) 0.4 (female)
    * 6 months to < 1 year: 0.5 (male) 0.5 (female)
    * 1 to < 2 years: 0.6 (male) 0.6 (female)
    * 2 to < 6 years: 0.8 (male) 0.8 (female)
    * 6 to < 10 years: 1 (male) 1 (female)
    * 10 to < 13 years: 1.2 (male) 1.2 (female)
    * 13 to < 16 years: 1.5 (male) 1.4 (female)
    * >= 16 years: 1.7 (male) 1.4 (female)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age (within 7 days prior to enrollment)
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 3 x ULN (=< 135 U/L) (within 7 days prior to enrollment) (for the purpose of this study, the ULN for SGPT is 45 U/L)
* Serum albumin >= 2 g/dL (within 7 days prior to enrollment)
* Shortening fraction of >= 27% by echocardiogram OR ejection fraction of >= 50% by multi-gated acquisition (MUGA)
* Corrected QT (by Bazett's formula [QTcB]) interval < 450 msecs
* Patients must be able to swallow tablets or liquid; use of a nasogastric or gastrostomy (G) tube is also allowed

Exclusion Criteria:

* Patients who are pregnant or breast-feeding are not eligible for this study as there is yet no available information regarding human fetal or teratogenic toxicities; negative pregnancy tests must be obtained in girls who are post-menarchal; patients of reproductive potential may not participate unless they have agreed to use an effective contraceptive method for the duration of study therapy; women of childbearing potential should be advised to use effective contraception for 4 months after the last dose of trametinib; trametinib may also potentially be secreted in milk and therefore breastfeeding women are excluded; female patients should not breastfeed during treatment with trametinib, and for 4 months following the last dose; male patients must use a condom during intercourse and agree not to father a child during therapy and for 4 months following discontinuation of trametinib to avoid unnecessary exposure of trametinib to the fetus
* Concomitant Medications

  * Corticosteroids: patients requiring corticosteroids who have not been on a stable or decreasing dose of corticosteroid for the 7 days prior to enrollment are not eligible; if used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid

    * Note: hydrocortisone used as a pre-medication to prevent transfusion related reactions is not considered a concomitant corticosteroid
  * Investigational drugs: patients who are currently receiving another investigational drug are not eligible
  * Anti-cancer agents: patients who are currently receiving other anti-cancer agents are not eligible (except patients receiving hydroxyurea, which may be continued until 24 hours prior to start of protocol therapy)
  * Anti-graft versus host disease (GVHD) or agents to prevent organ rejection post-transplant: patients who are receiving cyclosporine, tacrolimus or other agents to prevent either graft-versus-host disease post bone marrow transplant or organ rejection post-transplant are not eligible for this trial
  * Cardiac medications: any medications for treatment of left ventricular systolic dysfunction
* Patients who have an uncontrolled infection are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible
* Patients with a history of hepatic sinusoid obstructive syndrome (veno-occlusive disease) within the prior 3 months are not eligible
* Patients with a history of or current evidence/risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR) are not eligible
* Patients with a history of RVO or CSR, or predisposing factors to RVO or CSR (e.g., uncontrolled glaucoma or ocular hypertension
* Patients with uncontrolled systemic disease(s) such as hypertension or diabetes mellitus are not eligible; blood pressure must be =< the 95th percentile for age, height, and gender
* Patients with a history of allergic reaction attributed to compounds of similar chemical or biologic composition to the MEK inhibitor, trametinib are not eligible
* Patients with a clinical diagnosis of Noonan syndrome are not eligible; Note: patients with Casitas B-lineage lymphoma (CBL) syndrome, also known as Noonan-like syndrome, are eligible to enroll

Ages: 1 Month to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2018-09-09 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2026-10-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Stieglitz, Principal Investigator — Children's Oncology Group
Locations (57):
- United States (57):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Stieglitz E, Lee AG, Angus SP, Davis C, Barkauskas DA, Hall D, Kogan SC, Meyer J, Rhodes SD, Tasian SK, Xuei X, Shannon K, Loh ML, Fox E, Weigel BJ. Efficacy of the Allosteric MEK Inhibitor Trametinib in Relapsed and Refractory Juvenile Myelomonocytic Leukemia: a Report from the Children's Oncology Group. Cancer Discov. 2024 Sep 4;14(9):1590-1598. doi: 10.1158/2159-8290.CD-23-1376. PMID 38867349
- [Derived] McCullough KB, Kuhn AK, Patnaik MM. Treatment advances for pediatric and adult onset neoplasms with monocytosis. Curr Hematol Malig Rep. 2021 Jun;16(3):256-266. doi: 10.1007/s11899-021-00622-8. Epub 2021 Mar 16. PMID 33728588

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Trametinib)
Started | 10
Completed | 3
Not Completed | 7
Not completed — Physician Determines It Is In Patient's Best Interest | 4
Not completed — Progressive Disease | 3

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Trametinib)
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 1.96 [0.89 to 6.55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 1
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response
Description: Response rates will be calculated as the percent of evaluable patients who are responders, and confidence intervals will be constructed accounting for the two-stage design. A responder is defined as a patient who achieves a best response of PR or CR on the study prior to having an overall response of PD; all others will be considered non-responders. The definitions of response are based on a publication (PMID: 25552679) entitled "Criteria for evaluating response and outcome in clinical trials for children with juvenile myelomonocytic leukemia". Patients can be categorized as having experienced complete remission, partial remission, stable disease, or progressive disease based on a combination of clinical and molecular variables.
Time Frame: 12 cycles (1 cycle = 28 days)
Population: All patients who met the evaluable for response criteria outlined in section 9.4 of the ADVL1521 protocol.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Treatment (Trametinib)
Number analyzed (Participants) | 10
Percentage of patients | 50.0 [18.7 to 81.3]

2. Secondary Outcome: Incidence of Adverse Events
Description: Will be assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Will report the percentage of patients within each disease stratum who experienced a grade 3 or higher toxicity with attribution of possible, probable, or definite while on protocol therapy or within 30 days of the last dose of therapy.
Time Frame: Up to cycle 12 (1 cycle = 28 days)
Population: All patients who met the evaluable for response criteria outlined in section 9.4 of the ADVL1521 protocol.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Treatment (Trametinib)
Number analyzed (Participants) | 10
Percentage of patients | 30.0 [6.7 to 65.2]

3. Secondary Outcome: Pharmacokinetic (PK) Parameters of Trametinib
Description: A descriptive analysis of pharmacokinetic parameters of trametinib will be performed to define systemic exposure, drug clearance, Trametinib concentrations, and other pharmacokinetic parameters. The PK parameters will be summarized with simple summary statistics, including means, medians, ranges, and standard deviations (if numbers and distribution permit).
Time Frame: Up to cycle 12 (1 cycle = 28 days)
Population: Pharmacokinetic samples were collected and run, and the assay results were reviewed. However, two experts who reviewed the data found it to be uninterpretable because it was generated using incorrect standard curves.
Arm/Group | Treatment (Trametinib)
Number analyzed (Participants) | 0

4. Secondary Outcome: Trametinib Concentrations
Description: Will be measured by mass spectrometry. Will be analyzed descriptively. Values will be summarized with means and standard deviations.
Time Frame: Up to cycle 12 (1 cycle = 28 days)
Population: as for outcome 3
Arm/Group | Treatment (Trametinib)
Number analyzed (Participants) | 0

5. Secondary Outcome: Mutant Allele Burden
Description: Will be measured by next-generation sequencing. The percent change in mutant allele burden will be analyzed descriptively. Values will be summarized with means and standard deviations.
Time Frame: Up to cycle 12 (1 cycle = 28 days)
Population: All patients who met the evaluable for response criteria outlined in section 9.4 of the ADVL1521 protocol.
Measure: Mean (Standard Deviation); unit: Percent Change In Mutant Allele Burden
Arm/Group | Treatment (Trametinib)
Number analyzed (Participants) | 10
Percent Change In Mutant Allele Burden | 0.0 (0)

6. Secondary Outcome: Complete Response
Description: Complete Response rates will be calculated as the percent of evaluable patients who had an overall best response of Complete Response, and confidence intervals will be constructed accounting for the two-stage design.
Time Frame: 12 cycles (1 cycle = 28 days)
Population: All patients who met the evaluable for response criteria outlined in section 9.4 of the ADVL1521 protocol.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Treatment (Trametinib)
Number analyzed (Participants) | 10
Percentage of patients | 0.0 [0.0 to 30.8]

7. Secondary Outcome: Duration of Response
Description: Duration of response (Aim 1.2.5) will be defined as the time from first occurrence of PR or CR until the first occurrence of PD, death, or going off study. Patients who progress will be considered to have had an event, patients who die prior to progressing will be considered to have a competing event, and patients who go off study prior to progressing will be censored at time of last contact. The analysis will be done using the method of Gray.
Time Frame: Up to 5 years
Population: All patients who achieved an overall best response of Partial Response or Complete Response.
Measure: Median (Full Range); unit: years
Arm/Group | Treatment (Trametinib)
Number analyzed (Participants) | 5
years | 2.26 [0.87 to 2.78]

ADVERSE EVENTS:
Time Frame: Adverse Events monitored/assessed up to 30 days after treatment (12 cycles). All-Cause Mortality monitored/assessed up to 5 years from study enrollment.
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. All-Cause Mortality includes all deaths collected on the study. Ineligible patients are excluded from reporting of adverse events.
Arm/Group | Treatment (Trametinib)
All-Cause Mortality (participants affected / at risk) | 2/10
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Trametinib) (N=10)
Diarrhea (Gastrointestinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Sepsis (Infections and infestations) | 2
Stridor (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Trametinib) (N=10)
Anemia (Blood and lymphatic system disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1
Fever (General disorders) | 2
Folliculitis (Infections and infestations) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Neutrophil count decreased (Investigations) | 2
Paronychia (Infections and infestations) | 2
Platelet count decreased (Investigations) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Sinus tachycardia (Cardiac disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3
Urticaria (Skin and subcutaneous tissue disorders) | 1
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Soft tissue infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-22): https://cdn.clinicaltrials.gov/large-docs/15/NCT03190915/Prot_SAP_000.pdf